CLINICAL TRIAL: NCT00781027
Title: Fuchs' Endothelial Dystrophy and Cataract Surgery: Can Torsional Phacoemulsification Decrease the Risk for Corneal Decompensation
Brief Title: Fuchs' Torsional Phaco Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Dr. R.M.M.A. Nuijts, Department of Ophthalmology, University Hospital Maastricht
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MEC 08-2-081; NL24769.068.08
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2010-05

CONDITIONS: Fuchs' Endothelial Dystrophy; Phacoemulsification
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy | interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Torsional phacoemulsification
  Interventions: Procedure: Phacoemulsification
- 2 (Active Comparator): Longitudinal phacoemulsification
  Interventions: Procedure: Phacoemulsification

INTERVENTIONS:
Procedure: Phacoemulsification — Comparison of longitudinal phacoemulsification and torsional phacoemulsification

SUMMARY:
The primary objective is to compare the effect of torsional phacoemulsification and longitudinal phacoemulsification on central and peripheral corneal thickness/volume after cataract surgery in patients with Fuchs' endothelial dystrophy.

DETAILED DESCRIPTION:
Fuchs' endothelial dystrophy is a progressive, bilateral disease of the corneal endothelium, which eventually leads to corneal decompensation. In the early stage, some patients develop visually significant cataract. During cataract surgery ultrasound (US) power is used to emulsify the lens, which leads to endothelial cell loss and tissue damage. The reduction of US power has become the primary surgical goal in cataract surgery, which is especially important in patients with Fuchs' endothelial dystrophy to limit endothelial cell loss.

In 2006, Alcon Surgical introduced a torsional mode in its phacoemulsification system (Infiniti Vision System). It includes a handpiece that produces rotary oscillations of the phacoemulsification tip and is suggested to reduce the amount of US power required to remove the cataractous nucleus, because it does not produce repulsion and breaks up the cataract by shearing and not by the conventional jackhammer effect. This reduction in US power, could lead to less endothelial cell damage than the conventional (longitudinal) mode, which is reported recently for patients with hard cataract. It is important to investigate patients with Fuchs' endothelial dystrophy, because patients with a compromised endothelial cell layer will benefit the most from less endothelial cell damage. Consequently, this lower level of endothelial damage may postpone the date of keratoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Fuchs' endothelial dystrophy (all stages) and planning to undergo cataract surgery due to visually significant cataract
* Patients should be 40 years of age or older

Exclusion Criteria:

* Patients with Fuchs' dystrophy with a history of previous corneal or intraocular surgery
* Patients with a planned combined surgical procedure
* Patients who have other vision-affecting disorders than Fuchs' endothelial dystrophy

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change in central corneal thickness/corneal volume | 1, 7 days and 1 , 3 and 6 months postoperatively

SECONDARY OUTCOMES:
Changes in BCVA | 1, 7 days and 1, 3 and 6 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Rudy MMA Nuijts, MD, PhD, Study Director — Maastricht University Medical Center
Locations (1):
- University Hospital Maastricht, Maastricht, Netherlands

REFERENCES:
- [Derived] Doors M, Berendschot TT, Touwslager W, Webers CA, Nuijts RM. Phacopower modulation and the risk for postoperative corneal decompensation: a randomized clinical trial. JAMA Ophthalmol. 2013 Nov;131(11):1443-50. doi: 10.1001/jamaophthalmol.2013.5009. PMID 24030086